CLINICAL TRIAL: NCT04894435
Title: Immunogenicity and Adverse Events Following Immunization (AEFI) With Alternate Schedules of COVID-19 Vaccines in Canada: is "Mix and Match" of the Second Dose (MOSAIC-1;CT24a) and Additional Doses (MOSAIC-2 and MOSAIC-3;CT24b and CT24c) Safe and Immunogenic?
Brief Title: Mix and Match of the COVID-19 Vaccine for Safety and Immunogenicity
Acronym: MOSAIC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Immunization Research Network (Network)
Collaborators: Canadian Center for Vaccinology (Other); BC Children's Hospital Research Institute (Other); Children's Hospital Research Institute of Manitoba (Other); CHU de Quebec-Universite Laval (Other); Ottawa Hospital Research Institute (Other); Ontario Agency for Health Protection and Promotion (Other Government); University of Toronto (Other); Massachusetts General Hospital (Other); Interior Health (Industry); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CT24
Record Dates: First submitted 2021-05-18; First posted 2021-05-20 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; vaccine; clinical trial
MeSH Terms: conditions — COVID-19 | interventions — 2019-nCoV Vaccine mRNA-1273; BNT162 Vaccine; ChAdOx1 nCoV-19; Appointments and Schedules

STUDY DESIGN:
Intervention Model Description: M=Moderna SpikeVax mRNA; P=Pfizer/BioNTech Comirnaty mRNA; A=AstraZeneca Vaxzervia; C=Medicago Covifenz VLP
  MOSAIC 1:
  * Group 1 - M, M - 28 days
  * Group 2 - M, M - 112 days
  * Group 3 - M, P - 28 days
  * Group 4 - M, P - 112 days
  * Group 5 - P, P - 28 days
  * Group 6 - P, P - 112 days
  * Group 7 - P, M - 28 days
  * Group 8 - P, M - 112 days
  * Group 9 - A, M - 28 days
  * Group 10 - A, M - 112 days
  * Group 11 - A, P - 28 days
  * Group 12 - A, P - 112 days
  MOSAIC 2:
  * Group 1b - P, P, P
  * Group 2b - P, P, M
  * Group 3b - M, M, M
  * Group 4b - M, M, P
  * Group 5b - P and M in any order, M
  * Group 6b - P and M in any order, P
  * Group 7b - A, P or M, P
  * Group 8b - A, P or M, M
  * Group 9b - Any vaccine in any order, C (open-label)
  MOSAIC 3:
  * Group 1c - P, P, P, P
  * Group 2c - P, P, P, C
  * Group 3c - M, M, M, M
  * Group 4c - M, M, M, C
  * Group 5c - Any 3 in any order, P or M
  * Group 6c - Any 3 in any order, C
  * Group 7c - Any 3 in any order, C (open-label)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, laboratory staff, and statistical analysis personnel will be blinded to which vaccine they are receiving for those in randomized arms.
  Laboratory staff and statistical analysis personnel will be blinded to which vaccine they are receiving for those in open-label arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (28):
- Group 1: Moderna, Moderna - 28 Days apart (Active Comparator): Participants will be blinded and receive two doses (0.20 mg/mL each) of mRNA-1273 SARS-CoV-2 vaccine via intramuscular injection in the deltoid muscle 28 days apart.
  Vaccine-exposed participants will only be blinded to, and receive, the second injection.
  Interventions: Biological: mRNA-1273 SARS-CoV-2 vaccine; Other: 0, 28 day schedule
- Group 2: Moderna, Moderna - 112 days apart (Active Comparator): Participants will be blinded and receive two doses (0.20 mg/mL each) of mRNA-1273 SARS-CoV-2 vaccine at 0.20 mg/mL via intramuscular injection in the deltoid muscle 112 days apart.
  Vaccine-exposed participants will only be blinded to, and receive, the second injection.
  Interventions: Biological: mRNA-1273 SARS-CoV-2 vaccine; Other: 0, 112 day schedule
- Group 3: Moderna, Pfizer/BioNTech - 28 days apart (Active Comparator): Participants will be blinded and receive one dose (0.20 mg/mL) of mRNA-1273 SARS-CoV-2 vaccine via intramuscular injection in the deltoid muscle followed by one dose (0.3mL) of BNT162b2 vaccine after 28 days.
  Vaccine-exposed participants will only be blinded to, and receive, the second injection.
  Interventions: Biological: mRNA-1273 SARS-CoV-2 vaccine; Biological: BNT162b2; Other: 0, 28 day schedule
- Group 4: Moderna, Pfizer/BioNTech - 112 days apart (Active Comparator): Participants will be blinded and receive one dose (0.20 mg/mL) of mRNA-1273 SARS-CoV-2 vaccine via intramuscular injection in the deltoid muscle followed by one dose (0.3mL) of BNT162b2 vaccine after 112 days.
  Vaccine-exposed participants will only be blinded to, and receive, the second injection.
  Interventions: Biological: mRNA-1273 SARS-CoV-2 vaccine; Biological: BNT162b2; Other: 0, 112 day schedule
- Group 5: Pfizer/BioNTech, Pfizer/BioNTech - 28 days apart (Active Comparator): Participants will be blinded and receive two doses (0.3mL each) of BNT162b2 vaccine via intramuscular injection in the deltoid muscle 28 days apart.
  Vaccine-exposed participants will only be blinded to, and receive, the second injection.
  Interventions: Biological: BNT162b2; Other: 0, 28 day schedule
- Group 6: Pfizer/BioNTech, Pfizer/BioNTech - 112 days apart (Active Comparator): Participants will be blinded and receive two doses (0.3mL each) of BNT162b2 vaccine via intramuscular injection in the deltoid muscle 112 days apart.
  Vaccine-exposed participants will only be blinded to, and receive, the second injection.
  Interventions: Biological: BNT162b2; Other: 0, 112 day schedule
- Group 7: Pfizer/BioNTech, Moderna - 28 days apart (Active Comparator): Participants will be blinded and receive one dose (0.3mL) of BNT162b2 vaccine via intramuscular injection in the deltoid muscle followed by one dose (0.20 mg/mL) of mRNA-1273 SARS-CoV-2 vaccine after 28 days.
  Vaccine-exposed participants will only be blinded to, and receive, the second injection.
  Interventions: Biological: mRNA-1273 SARS-CoV-2 vaccine; Biological: BNT162b2; Other: 0, 28 day schedule
- Group 8: Pfizer/BioNTech, Moderna - 112 days apart (Active Comparator): Participants will be blinded and receive one dose (0.3mL) of BNT162b2 vaccine via intramuscular injection in the deltoid muscle followed by one dose (0.20 mg/mL) of mRNA-1273 SARS-CoV-2 vaccine after 112 days.
  Vaccine-exposed participants will only be blinded to, and receive, the second injection.
  Interventions: Biological: mRNA-1273 SARS-CoV-2 vaccine; Biological: BNT162b2; Other: 0, 112 day schedule
- Group 9: Astra Zeneca, Moderna - 28 days apart (Active Comparator): Participants will be blinded and receive one dose (0.5 ml) of ChAdOx1-S [recombinant] vaccine via intramuscular injection in the deltoid muscle followed by one dose (0.20 mg/mL) of mRNA-1273 SARS-CoV-2 vaccine after 28 days.
  Vaccine-exposed participants will only be blinded to, and receive, the second injection.
  Interventions: Biological: mRNA-1273 SARS-CoV-2 vaccine; Biological: ChAdOx1-S [recombinant]; Other: 0, 28 day schedule
- Group 10: Astra Zeneca, Moderna - 112 days apart (Active Comparator): Participants will be blinded and receive one dose (0.5 ml) of ChAdOx1-S [recombinant] vaccine via intramuscular injection in the deltoid muscle followed by one dose (0.20 mg/mL) of mRNA-1273 SARS-CoV-2 vaccine after 112 days.
  Vaccine-exposed participants will only be blinded to, and receive, the second injection.
  Interventions: Biological: mRNA-1273 SARS-CoV-2 vaccine; Biological: ChAdOx1-S [recombinant]; Other: 0, 112 day schedule
- Group 11: Astra Zeneca, Pfizer/BioNTech - 28 days apart (Active Comparator): Participants will be blinded and receive one dose (0.5 ml) of ChAdOx1-S [recombinant] vaccine via intramuscular injection in the deltoid muscle followed by one dose (0.3 mL) of BNT162b2 vaccine after 28 days.
  Vaccine-exposed participants will only be blinded to, and receive, the second injection.
  Interventions: Biological: BNT162b2; Biological: ChAdOx1-S [recombinant]; Other: 0, 28 day schedule
- Group 12: Astra Zeneca, Pfizer/BioNTech - 112 days apart (Active Comparator): Participants will be blinded and receive one dose (0.5 ml) of ChAdOx1-S [recombinant] vaccine via intramuscular injection in the deltoid muscle followed by one dose (0.3 mL) of BNT162b2 vaccine after 112 days.
  Vaccine-exposed participants will only be blinded to, and receive, the second injection.
  Interventions: Biological: BNT162b2; Biological: ChAdOx1-S [recombinant]; Other: 0, 112 day schedule
- Group 1b (Active Comparator): Participants will be blinded and receive one dose (0.3mL) of BNT162b2 vaccine via intramuscular injection in the deltoid muscle.
  Interventions: Biological: BNT162b2
- Group 2b (Active Comparator): Participants will be blinded and receive one half dose (0.25mL) of mRNA-1273 vaccine via intramuscular injection in the deltoid muscle.
  Interventions: Biological: mRNA-1273 SARS-CoV-2 vaccine
- Group 3b (Active Comparator): Participants will be blinded and receive one half dose (0.25mL) of mRNA-1273 vaccine via intramuscular injection in the deltoid muscle.
  Interventions: Biological: mRNA-1273 SARS-CoV-2 vaccine
- Group 4b (Active Comparator): Participants will be blinded and receive one dose (0.3mL) of BNT162b2 vaccine via intramuscular injection in the deltoid muscle.
  Interventions: Biological: BNT162b2
- Group 5b (Active Comparator): Participants will be blinded and receive one half dose (0.25mL) of mRNA-1273 vaccine via intramuscular injection in the deltoid muscle.
  Interventions: Biological: mRNA-1273 SARS-CoV-2 vaccine
- Group 6b (Active Comparator): Participants will be blinded and receive one dose (0.3mL) of BNT162b2 vaccine via intramuscular injection in the deltoid muscle.
  Interventions: Biological: BNT162b2
- Group 7b (Active Comparator): Participants will be blinded and receive one dose (0.3mL) of BNT162b2 vaccine via intramuscular injection in the deltoid muscle.
  Interventions: Biological: BNT162b2
- Group 8b (Active Comparator): Participants will be blinded and receive one half dose (0.25mL) of mRNA-1273 vaccine via intramuscular injection in the deltoid muscle.
  Interventions: Biological: mRNA-1273 SARS-CoV-2 vaccine
- Group 9b (Experimental): Participants will receive one dose (0.5mL) of Covifenz vaccine via intramuscular injection in the deltoid muscle.
  Interventions: Biological: Covifenz
- Group 1c (Active Comparator): Participants will be blinded and receive one dose (0.3mL) of BNT162b2 vaccine via intramuscular injection in the deltoid muscle.
  Interventions: Biological: BNT162b2
- Group 2c (Active Comparator): Participants will be blinded and receive one dose (0.5mL) of Covifenz vaccine via intramuscular injection in the deltoid muscle.
  Interventions: Biological: Covifenz
- Group 3c (Active Comparator): Participants will be blinded and receive one half dose (0.25mL) of mRNA-1273 vaccine via intramuscular injection in the deltoid muscle.
  Interventions: Biological: mRNA-1273 SARS-CoV-2 vaccine
- Group 4c (Active Comparator): Participants will be blinded and receive one dose (0.5mL) of Covifenz vaccine via intramuscular injection in the deltoid muscle.
  Interventions: Biological: Covifenz
- Group 5c (Active Comparator): Participants will be blinded and receive either one dose (0.3mL) of BNT162b2 or one half dose (0.25mL) of mRNA-1273 via intramuscular injection in the deltoid muscle.
  Interventions: Biological: mRNA-1273 SARS-CoV-2 vaccine; Biological: BNT162b2
- Group 6c (Active Comparator): Participants will be blinded and receive one dose (0.5mL) of Covifenz vaccine via intramuscular injection in the deltoid muscle.
  Interventions: Biological: Covifenz
- Group 7c (Experimental): Participants will receive one dose (0.5mL) of Covifenz vaccine via intramuscular injection in the deltoid muscle.
  Interventions: Biological: Covifenz

INTERVENTIONS:
Biological: mRNA-1273 SARS-CoV-2 vaccine — Contains 1.26 mg of CX-024414 mRNA and 24.38 mg of SM-102 LNP as a white to off-white dispersion in preservative-free diluent buffer at pH 7.5.
  Other Names: COVID-19 Vaccine Moderna; Spikevax
  Arms: Group 10: Astra Zeneca, Moderna - 112 days apart; Group 1: Moderna, Moderna - 28 Days apart; Group 2: Moderna, Moderna - 112 days apart; Group 2b; Group 3: Moderna, Pfizer/BioNTech - 28 days apart; Group 3b; Group 3c; Group 4: Moderna, Pfizer/BioNTech - 112 days apart; Group 5b; Group 5c; Group 7: Pfizer/BioNTech, Moderna - 28 days apart; Group 8: Pfizer/BioNTech, Moderna - 112 days apart; Group 8b; Group 9: Astra Zeneca, Moderna - 28 days apart
Biological: BNT162b2 — A white to off-white, sterile, preservative-free, frozen suspension for intramuscular injection, supplied with 0.9% sodium chloride diluent for injection plastic ampoules.
  Other Names: Pfizer-BioNTech COVID-19 Vaccine; Comirnaty
  Arms: Group 11: Astra Zeneca, Pfizer/BioNTech - 28 days apart; Group 12: Astra Zeneca, Pfizer/BioNTech - 112 days apart; Group 1b; Group 1c; Group 3: Moderna, Pfizer/BioNTech - 28 days apart; Group 4: Moderna, Pfizer/BioNTech - 112 days apart; Group 4b; Group 5: Pfizer/BioNTech, Pfizer/BioNTech - 28 days apart; Group 5c; Group 6: Pfizer/BioNTech, Pfizer/BioNTech - 112 days apart; Group 6b; Group 7: Pfizer/BioNTech, Moderna - 28 days apart; Group 7b; Group 8: Pfizer/BioNTech, Moderna - 112 days apart
Biological: ChAdOx1-S [recombinant] — A colourless to slightly brown, clear to slightly opaque solution containing 5 x 1010 viral particles (not less than 2.5 x 108 infectious units).
  Other Names: Astra Zeneca COVID-19 Vaccine; COVISHIELD AstraZeneca COVID-19 Vaccine; Vaxzevria
  Arms: Group 10: Astra Zeneca, Moderna - 112 days apart; Group 11: Astra Zeneca, Pfizer/BioNTech - 28 days apart; Group 12: Astra Zeneca, Pfizer/BioNTech - 112 days apart; Group 9: Astra Zeneca, Moderna - 28 days apart
Other: 0, 28 day schedule — Second injection administered 28 days post first injection
  Arms: Group 11: Astra Zeneca, Pfizer/BioNTech - 28 days apart; Group 1: Moderna, Moderna - 28 Days apart; Group 3: Moderna, Pfizer/BioNTech - 28 days apart; Group 5: Pfizer/BioNTech, Pfizer/BioNTech - 28 days apart; Group 7: Pfizer/BioNTech, Moderna - 28 days apart; Group 9: Astra Zeneca, Moderna - 28 days apart
Other: 0, 112 day schedule — Second injection administered 112 days post first injection
  Arms: Group 10: Astra Zeneca, Moderna - 112 days apart; Group 12: Astra Zeneca, Pfizer/BioNTech - 112 days apart; Group 2: Moderna, Moderna - 112 days apart; Group 4: Moderna, Pfizer/BioNTech - 112 days apart; Group 6: Pfizer/BioNTech, Pfizer/BioNTech - 112 days apart; Group 8: Pfizer/BioNTech, Moderna - 112 days apart
Biological: Covifenz — COVIFENZ is an emulsion for intramuscular injection. The 3.75 mcg antigen component of COVIFENZ is a suspension, which must be mixed 1:1 with the 0.25 mL AS03 adjuvant emulsion component prior to administration
  Other Names: Medicago COVID-19 vaccine
  Arms: Group 2c; Group 4c; Group 6c; Group 7c; Group 9b

SUMMARY:
The main goals of this study are to assess the immune response and safety of two different vaccines for first, second, third and fourth doses as well as for differing intervals between the first and second dose of two-dose vaccines.

DETAILED DESCRIPTION:
For dose 1 and 2, the currently available mRNA vaccines (Pfizer-BioNTech BNT162b2 and Moderna mRNA-1273) are two dose vaccines which were studied in schedules of either 0 and 21 days or 0 and 28 days, respectively. The ChAdOx1 nCOV-19 (Astra-Zeneca) adenovirus-vectored vaccine is authorized to be given in two doses one month to 12 weeks apart. We will compare the interval 0, 28 days to a 0, 112 days (16 weeks) schedule, and assess the immunogenicity of both heterogeneous and heterologous second doses using the Canadian schedule.

For dose 3, the currently available mRNA vaccines (Pfizer-BioNTech BNT162b2 and Moderna mRNA-1273) and plant-based virus-like particle (Medicago Covifenz) are anticipated to be administered 6 months apart. We will assess the immunogenicity of both heterogeneous and heterologous third doses using the Canadian schedule.

For dose 4, the currently available mRNA vaccines (Pfizer-BioNTech BNT162b2 and Moderna mRNA-1273) and plant-based virus-like particle (Medicago Covifenz) are anticipated to be administered 3 months apart. We will assess the immunogenicity of both heterogeneous and heterologous third doses using the Canadian schedule.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is willing and able to give written informed consent to participate in the study
2. Age 18 years of age or older in good health or with mild or moderate stable co-morbidities at the time of enrolment
3. Able and willing to complete all the scheduled study procedures during the whole study follow-up period
4. If female of child-bearing potential and heterosexually active, has practiced adequate contraception for 30 days prior to injection, has a negative pregnancy test on the day of injection, and has agreed to continue adequate contraception until 3 months after the final dose of study vaccine (Please refer to the definition section for a description of child-bearing potential and adequate contraception)
5. MOSAIC-1 Vaccine-exposed subgroups: have received or are booked to receive the first dose of an authorized COVID-19 vaccine in the 55 days prior to Visit 1 (documentation of receipt required)
6. MOSAIC -1 Vaccine naïve subgroups: have not received an authorized COVID-19 vaccine at any time
7. MOSAIC-2 participants have received two doses of COVID-19 vaccines authorized in Canada ≥6 months prior to study vaccine administration (documentation of receipt required)
8. MOSAIC-3 participants have received three doses of COVID-19 vaccines authorized in Canada ≥3 months prior to study vaccine administration (documentation of receipt required)

Exclusion Criteria:

1. Inability or unwillingness of participant or legally acceptable representative to give written informed consent
2. Any confirmed or suspected immunosuppressive or immunodeficient state; asplenia, or immunosuppressant medication within the past 6 months except short term oral steroids (≤14 days duration) or topical steroids
3. Current diagnosis or treatment for cancer (except basal cell carcinoma of the skin)
4. Administration of immunoglobulins and/or any blood products within 3 months preceding the first dose of study vaccine and for one month after the last dose of study vaccine
5. Allergy to any study vaccine or any active substance in a study vaccine
6. Bleeding disorder or history of significant bleeding following IM injections or venipuncture
7. Continuous use of anticoagulants
8. A history of anaphylaxis to a previous vaccine
9. Pregnancy or intent to become pregnant during the study or within 3 months of the last dose of study vaccine
10. MOSAIC-1: History of laboratory-confirmed COVID-19 disease prior to enrolment by participant report
11. Administration of a live virus vaccine within 4 weeks prior to study vaccine receipt.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 669 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Antibody response to SARS-CoV-2 S protein after 2 doses | Day 56
  The co-primary outcome for the non-inferiority comparison of 0, 28-day schedules with heterologous second dose is the immune response to SARS-CoV-2 at day 56 (28 days after the second dose of vaccine) based on anti-spike antibody titers.
Antibody response to SARS-CoV-2 S protein after 2 doses | Day 140
  The co-primary outcome for the non-inferiority comparison of schedules in which the timing of the second dose of vaccine is different (0, 28 days v 0, 112 days) is the immune response to SARS-CoV-2 at day 140 (28 days after the last dose in the 0, 112 day schedule) based on anti-spike antibody titers.
Antibody response to SARS-CoV-2 S protein after 3 doses | Day 28
  To determine if a vaccination schedule with a heterologous third dose of a COVID-19 vaccine induces a non-inferior serum immune response to SARS-CoV-2, compared to a third dose/booster with a homologous vaccine.
Antibody response to SARS-CoV-2 S protein after 4 doses | Day 28
  To determine if a vaccination schedule with a heterologous fourth dose of a COVID-19 vaccine induces a non-inferior serum immune response to SARS-CoV-2, compared to a third dose/booster with a homologous vaccine.

SECONDARY OUTCOMES:
Durability of antibody response to SARS-CoV-2 S over 12 months after 2 doses | Baseline and Days 28, 56, 112, 140, 365
  Assess durability of immune responses in each study group over 12 months based on anti-spike antibody titers and pseudoneutralization assay.
Pseudoneutralization assay, T cell testing, Antibody dependent cellular cytotoxicity (ADCC), Antibody avidity, RNA seq after 2 doses | Days 28, 56, 112, 140, 365
  Characterization of the immune response to COVID-19 vaccines in schedules with 0, 28 days versus 0, 112 days dosing and heterologous schedules to day 365.
Incidence of grade 3 solicited local and systemic adverse events, SAEs, AEFIs, MAAEs, AESIs in the 7 days following vaccine receipt after 2 doses | From time of first study injection through Day 365.
  Description of safety outcomes over 12 months post-vaccination including SAEs (serious adverse events), provincially reportable AEFIs (adverse events following immunization), MAAEs (medically attended adverse events), AESIs (adverse events of special interest).
Incidence of grade 3 solicited local and systemic adverse events, SAEs, AEFIs, MAAEs, AESIs in the 7 days following vaccine receipt after 3 doses | From time of first study injection through Day 365.
  Description of safety outcomes over 12 months post-vaccination including SAEs (serious adverse events), provincially reportable AEFIs (adverse events following immunization), MAAEs (medically attended adverse events), AESIs (adverse events of special interest).
Acceptability of vaccines as determined by participant-completed questionnaire after 2 doses | Days 56, 140, and 365
  Four 5 point likert scale type questions asking whether they would want to receive the vaccine again, recommend it to a friend, whether they were anxious about receiving it, and whether they would prefer a more painful injection if it conferred better protection.
Acceptability of vaccines as determined by participant-completed questionnaire after 3 doses | Days 28, 180
  Four 5 point likert scale type questions asking whether they would want to receive the vaccine again, recommend it to a friend, whether they were anxious about receiving it, and whether they would prefer a more painful injection if it conferred better protection.
Antibody to SARS-CoV-2 S and N, RBD after 3 doses | Days 180 and 365
  Assess durability of the immune responses in each study group over 12 months after the study vaccine.
Pseudoneutralization assay, T cell testing, Antibody dependent cellular cytotoxicity after 3 doses | Day 365
  Further characterize the immune response to COVID-19 vaccine in schedules with homologous and heterologous third doses to day 365
Incidence of grade 3 solicited local and systemic adverse events, SAEs, AEFIs, MAAEs, AESIs in the 7 days following vaccine receipt after 4 doses | From time of first study injection through Day 365.
  Description of safety outcomes over 12 months post-vaccination including SAEs (serious adverse events), provincially reportable AEFIs (adverse events following immunization), MAAEs (medically attended adverse events), AESIs (adverse events of special interest).
Acceptability of vaccines as determined by participant-completed questionnaire after 4 doses | Days 28, 180
  Four 5 point likert scale type questions asking whether they would want to receive the vaccine again(Yes, definitely; Yes, probably; I don't know; No, probably not; No, definitely not), recommend it to a friend(Yes, definitely; Yes, probably; I don't know; No, probably not; No, definitely not), whether they were anxious about receiving it(Not at all; A little; Moderately; Very; Extremely), and whether they would prefer a more painful injection if it conferred better protection(Vaccine A; Vaccine B; No preference; Unsure/don't know).
Antibody to SARS-CoV-2 S and N, RBD after 4 doses | Days 180 and 365
  Assess durability of the immune responses in each study group over 12 months after the study vaccine.
Antibody dependent cellular cytotoxicity after 4 doses | Day 365
  Further characterize the immune response to COVID-19 vaccine in schedules with homologous and heterologous third doses to day 365
Pseudoneutralization assay after 4 doses | Day 365
  Measuring the 50% Neutralization Titer to further characterize the immune response to COVID-19 vaccine in schedules with homologous and heterologous third doses to day 365
T cell testing after 4 doses | Day 365
  Measuring the number of T cells to further characterize the immune response to COVID-19 vaccine in schedules with homologous and heterologous third doses to day 365

OTHER OUTCOMES:
Exploratory assessment of interval between dose 1 and 2 on immune response after 3 or 4 doses | From time of first study injection through Day 365.
  Assess the role of intervals between first and second doses of the primary immunization schedule, and between 2nd and 3rd doses, on immune responses after the third dose over the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Langley, Principal Investigator — Dalhousie University/CIRN
Locations (8):
- Canada (8):
  - Royal Inland Hospital, Kamloops, British Columbia
  - Penticton Regional Hospital, Penticton, British Columbia
  - BC Children's Hospital Research Institute, Vancouver, British Columbia
  - Children's Hospital Research Institute of Manitoba, Winnipeg, Manitoba
  - Canadian Center for Vaccinology, Halifax, Nova Scotia
  - Ottawa Hospital Research Institute, University of Ottawa, Ottawa, Ontario
  - McGill University Health Centre Vaccine Study Centre, Montreal, Quebec
  - CHU de Québec, Université Laval, Québec, Quebec